CLINICAL TRIAL: NCT03251053
Title: Adverse Airway Effects of Inhaled Nicotine From Tobacco and E-Cigarettes
Brief Title: Adverse Airway Effects From Tobacco and E-Cigarettes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Miami VA Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Campos, MD, Miami VA Healthcare System
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 1251.09
Record Dates: First submitted 2017-07-25; First posted 2017-08-16 (Actual); Last update posted 2017-08-16 (Actual); Status verified 2017-08

CONDITIONS: Airway Morbidity; Smoking Cessation; Nicotine Adverse Reaction; Smoking, Tobacco; Smoking, Cigarette
MeSH Terms: conditions — Smoking Cessation; Tobacco Smoking; Cigarette Smoking

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Electronic cigarette use (Experimental): Subjects who try to switch to electronic cigarettes (EC) and subjects who successfully switch to EC.
  Interventions: Device: Electronic cigarette use
- Control regular cigarette smokers (Other): Habitual smokers without EC use
  Interventions: Device: Electronic cigarette use; Other: Control regular cigarette smokers

INTERVENTIONS:
Device: Electronic cigarette use — Replacement of tobacco smoking with electronic cigarette vaping
Other: Control regular cigarette smokers
  Arms: Control regular cigarette smokers

SUMMARY:
The purpose of the study conducted at VA Medical Center in Miami is to determine if smoking electronic cigarettes (known as e-cigarettes) that contain nicotine have less negative effects than regular cigarettes on the person's respiratory health. We will assess this by measuring pulmonary function tests, several body molecules and functionality of the airway cells. We will also evaluate how smokers can maintain exclusive electronic cigarettes use.

In this study, some people will continue to smoke regular tobacco cigarettes while others will switch to a nicotine-containing electronic cigarette.

DETAILED DESCRIPTION:
The study will evaluate the airway epithelial effects of EC (electronic cigarettes) vapor containing nicotine when used as a tobacco replacement tool. By using active cigarette smokers as a comparator group, the study will increase our knowledge of whether the use of ECs is more or less harmful than continuation of tobacco smoking. This study will examine the in vivo effects of EC vapors in nasal ion transport and TGF-β levels as well as in serum inflammatory biomarkers.

As the primary endpoint, nasal ion transport will be assessed by nasal potential difference (NPD), which measures the voltage potential resulting from epithelial ion fluxes at the mucosal surface in vivo. Ion transport across nasal epithelia is representative for findings in distal airways. Since NPD directly measures the changes in ion transport expected to influence mucociliary clearance (MCC) and therefore overall outcome and since changes of NPD measurements are indirectly linked to lung function changes and MCC in trials with cystic fibrosis patients, we believe that NPD lends itself as a reasonable surrogate for MCC for this clinical trial.

As secondary endpoints, we will also measure TGF-ß levels in nasal secretions and expression in nasal cells to correlate these with the level of CFTR and CaCC-mediated Cl- conductance (CFTR is known to show decreased function with elevated TGF-β). In addition plasma samples will be collected to study systemic markers of inflammation as well as toxic substances that may result from vaping and smoking.

The design is a smoking replacement trial, in which we will compare changes in upper airway ion transport and inflammation in smokers who switch to EC vaping versus subjects that continue to smoke tobacco cigarettes. In addition, we will use the trial design to evaluate the feasibility of using the EC as a means to quit tobacco use.

The study will last up to16 weeks with weekly visits. Subjects must replace completely cigarettes with EC within the first 4 visits (week 4) and maintain exclusive use for the following 12 visits. Adherence is asses with exhaled carbon monoxide and/or carboxyhemoglobin when needed. The study involves scheduled blood draws for research samples.

There will be total of 16 visits to the study clinic. Besides blood draws and NPD, the study will include questionnaires, lung function testing and adverse event recording.

ELIGIBILITY:
Inclusion Criteria:

* Subjects that actively smoke and have a history of at least 5 pack-years

Exclusion Criteria:

* HIV,marijuana use, asthma and other concomitant inflammatory pulmonary disorders, subjects with known pulmonary diseases including malignancies, subjects with prior thoracic surgery and subjects that used oral corticosteroids or antibiotics within the prior 3 months, subjects with allergies to study medications and subjects incapable of providing informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2021-03-28 (Estimated); Study Completion 2021-03-28 (Estimated)

PRIMARY OUTCOMES:
Change in nasal potential difference (NPD) | 11 weeks of transitioning
  nasal potential difference (NPD) before and after replacing tobacco cigarettes with electronic cigarettes

SECONDARY OUTCOMES:
change in Inflammatory markers smoking to electronic cigarettes | 11 weeks of transitioning
  TGF-ß levels in nasal secretions before and after replacing tobacco cigarettes with electronic cigarettes

CONTACTS AND LOCATIONS:
Overall Officials: Michael Campos, Principal Investigator — Miami VA Healthcare System
Locations (1):
- Miami VA Healthcare System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No